CLINICAL TRIAL: NCT06062485
Title: Efficacy and Safety of Surufatinib Combined With Toripalimab and AG Regiments for First-line Treatment of Unresectable or Relapsing Metastatic Ampullary Carcinoma
Brief Title: Surufatinib Combined With Toripalimab and AG Regiments for First-line Treatment of Unresectable or Relapsing Metastatic Ampullary Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-E2-BTC-101
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-04

CONDITIONS: Ampullary Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: Surufatinib+Toripalimab+AG

INTERVENTIONS:
Drug: Surufatinib+Toripalimab+AG — This is a single-arm, prospective, exploratory clinical study of unresectable or relapsing metastatic ampullary tumors who were not systematically treated with surufatinib in combination with PD-1 antibody and AG regimen.Until the investigator assesses loss of clinical benefit, unacceptable toxicity, decision by the investigator or subject to withdraw treatment, or death, whichever comes first.The AG regimen does not exceed 8 cycles, and maintenance therapy with surufatinib combined with toripalimab can be continued if the patient has not progressed after 8 cycles. The treatment period was 21 days; Tumor treatment and survival status were recorded until disease progression (RECIST 1.1) or death (during patient treatment).
  Surufatinib (200mg，qd，Q3W）；Toripalimab(240mg IV d1, Q3W)；AG（Albumin-bound paclitaxel: 125mg/m2，IV，d1，d8，Q3W）Gemcitabine: 1000 mg/m2, IV，d1，d8，Q3W）

SUMMARY:
A Phase Ⅱ, single-arm study to assess the safety, tolerability, and efficacy of Surufatinib Combination With Toripalimab in Patients With recurrent or metastatic ampulla tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old;
2. Unresectable or relapses metastatic ampullary malignancies identified by histopathology or cytology,with histological subtypes of parenteral type;
3. Have not received systematic treatment for unresectable or metastatic ampulla malignant tumor;A scheme of adjuvant or neoadjuvant chemotherapy and 6 months after the chemotherapy recurrence can into the group;
4. ECOG score 0 or 1;
5. Expected survival≥12 weeks;
6. Have at least one measurable lesion;
7. Major organ functions within 7 days prior to treatment shall meet the following criteria:

(1)Hemoglobin(HB)≥90 g/L; (2)neutrophil absolute value(ANC)≥1.5×109/L; (3)Platelet(PLT)≥100×109/L;

8.Biochemical examination shall meet the following standards:

1. Total bilirubin(TBIL)≤3 times the upper limit of normal value(ULN);
2. ALT and aspartate aminotransferase AST≤2.5×ULN,and ALT and AST≤5×ULN with liver metastasis;
3. Serum creatinine(Cr)≤1.5×ULN or creatinine clearance(CCr)≥60ml/min;

9.Doppler ultrasound evaluation:left ventricular ejection fraction(LVEF)≥the lower limit of normal value(50%)；

10.Patients of reproductive age(including female and male patients'female companions)must use effective birth control measures;

11.Subjects voluntarily joined the study and signed an informed consent form(ICF);

12.It is expected that the patient has good compliance and can follow up the efficacy and adverse reactions according to the protocol requirements.

Exclusion Criteria:

1. Patients who have previously been treated with small-molecule drugs similar to VEGFR-TKI,such as Anlotinib,Sunitinib,Sorafenib,Lenvatinib,Apatinib,etc.
2. Anti-pd-1 or anti-PD-L1/L2 antibodies or anti-cytotoxic T lymphocyte-associated antigen(CTLA-4)antibodies were used in the past;
3. Malignant ampulla obstruction after clinical intervention was not resolved or anti-infective therapy was required 14 days before the first study of drug therapy;
4. Patients with severe allergic history or allergic constitution;
5. Pregnant or lactating women;
6. Patients who have participated in other clinical trials and have not terminated the trials;
7. Patients with any severe and/or uncontrolled medical condition,including:

(1)Patients with unsatisfactory blood pressure control(systolic blood pressure≥150 mmHg,diastolic blood pressure≥100 mmHg); (2)Patients with grade I or above myocardial ischemia or myocardial infarction,arrhythmias(including QTc≥480ms),and≥grade 2 congestive heart failure(New York Heart Association(NYHA)grades); (3)Active or uncontrolled severe infection(≥CTC AE grade 2 infection); (4)Cirrhosis,decompensated liver disease,active hepatitis or chronic hepatitis require antiviral therapy; (5)Renal failure requiring hemodialysis or peritoneal dialysis; (6)A history of immunodeficiency,including HIV positive or other acquired or congenital immunodeficiency diseases,or a history of organ transplantation; (7)Urine protein≥++was indicated by two consecutive urine routine,and the 24-hour urine protein quantity was confirmed to be>1.0 g; (8)Mental illness,including epilepsy,dementia,severe depression,mania,etc.

8.Received major surgical treatment,open biopsy,or significant traumatic injury within 28 days prior to grouping(specifically in conjunction with clinical evaluation);

9.History of any active autoimmune disease or autoimmune disease,including but not limited to interstitial pneumonia,uveitis,inflammatory bowel disease,hepatitis,pituitary inflammation,vasculitis,systemic lupus erythematosus,etc.;

10.The patient currently has active gastric and duodenal ulcers,ulcerative colitis and other digestive diseases,or active bleeding from unexcised tumors,or other conditions determined by researchers that may cause gastrointestinal bleeding and perforation;

11.Patients with any physical signs or history of bleeding,regardless of severity;Unhealed wounds,ulcers,or fractures were observed in patients with any bleeding or bleeding events≥CTCAE grade 3 during the first 4 weeks of enrollment;

12.Experienced arteriovenous thrombotic events,such as cerebrovascular accidents(including temporary ischemic attacks),deep vein thrombosis and pulmonary embolism,within 6 months;

13.Those who have a history of psychotropic substance abuse and cannot abstain or have mental disorders;

14.Subjects with dysphagia or known drug absorption disorders.

15.The researchers considered other conditions unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1

SECONDARY OUTCOMES:
Progression free survival (PFS) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks, until the occurrence of progressive disease (PD), using RECIST v 1.1
Overall survival (OS） | from randomization until death due to any cause, assessed up to 3 year
  Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Disease control rate (DCR） | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Safety and tolerance evaluated by incidence, severity and outcomes of AEs | from first dose to 30 days post the last dose
  Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 5.0

IPD SHARING:
Plan to Share IPD: Undecided